CLINICAL TRIAL: NCT00309933
Title: Quality of Life in Younger Breast Cancer Survivors
Brief Title: Quality of Life in Female Breast Cancer Survivors and Their Spouse, Partner, or Acquaintance
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000460234; ECOG-E2Z04
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Cancer Survivor; Cognitive/Functional Effects; Psychosocial Effects of Cancer and Its Treatment; Sexuality and Reproductive Issues; Spiritual Concerns
Keywords: cognitive/functional effects; spiritual concerns; sexuality and reproductive issues; psychosocial effects of cancer and its treatment; cancer survivor; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Sexuality | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cognitive assessment
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying quality of life in breast cancer survivors may help determine the long-term effects of breast cancer and may help improve the quality of life for future breast cancer survivors.

PURPOSE: This clinical trial is studying quality of life in female breast cancer survivors and their spouse, partner, or acquaintance.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the quality of life (physical functioning, psychological functioning, social functioning, and spiritual functioning) of female breast cancer survivors who were age 45 or younger at the time of diagnosis with the quality of life of female breast cancer survivors who were age 55 to 70 at time of diagnosis (considering type of surgical treatment [lumpectomy vs mastectomy], hormonal treatments, and time since diagnosis as covariates) and age-matched (to the younger group) females with no history of breast cancer.
* Compare the quality of life (physical functioning, psychological functioning, social functioning, and spiritual functioning) of partners of breast cancer survivors who were age 45 or younger at time of diagnosis with the quality of life of partners of breast cancer survivors who were age 55 to 70 at diagnosis and partners of age-matched (to the younger group) females with no history of breast cancer.
* Test and compare quality of life models that identify the variables that mediate between antecedent variables of personal characteristics, diagnostic and treatment characteristics, and quality of life outcomes in order to determine where interventions to improve quality of life should be targeted.
* Explore the relationship of partner antecedent, mediating, and outcome variables as predictors or mediators of outcome variables for breast cancer survivors.

OUTLINE: This is a multicenter study.

Patients, spouse or partner of patients, age-matched acquaintances of patients, and partner of acquaintances complete questionnaires over 60-90 minutes about personal characteristics, self-efficacy, coping, social support, health care provider communication, physical, psychological, social, and spiritual functioning, and quality of life. After completing the study questionnaires, patients and age-matched acquaintances of patients are interviewed via telephone over 30 minutes for cognitive function assessment. A random subset of patients and spouses/partners of patients are interviewed via telephone over 45-60 minutes, using data-generating and open-ended questions, regarding physical functioning, sexual and reproductive issues, psychological issues, social impact, and methods used to deal with breast cancer survivor concerns.

Disease and treatment characteristics of patients are obtained from medical records.

PROJECTED ACCRUAL: A total of 2,697 patients, spouse or partner of patients, age-matched female acquaintances of patients, and partner of acquaintances will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient

  * Female breast cancer survivor with age at initial diagnosis in 1 of the following ranges:

    * 18 to 45
    * 55 to 78
  * Must have enrolled and participated in ECOG study CLB-9741, E-1199, or E-2197
  * Must have received chemotherapy at least 3 years, but no more than 8 years prior to this study entry
  * Disease free at the time of this study entry
* Spouse or partner of the patient, age-matched female acquaintances of the patient (in the younger patient group), or partner of acquaintances

  * Spouse or partner of the patient may be either gender
  * Age-matched female acquaintance is defined as within 5 years of age difference of the patient in younger group (18-45 years of age)

    * With a similar level of education and race of the patient
    * Not a personal friend of the patient
    * No history of breast cancer

PATIENT CHARACTERISTICS:

* Must reside in the continental U.S. and speak English (for patients)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2697 (Estimated)
Dates: Start 2006-04-03 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the quality of life
Comparison of the quality of life of partners
Comparison of quality of life models
Correlation between partner antecedent, mediating, and outcome variables with patient outcome variables

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Champion, DNS, Study Chair — Indiana University Melvin and Bren Simon Cancer Center; George W. Sledge, MD — Indiana University Melvin and Bren Simon Cancer Center; Lynne Wagner, MD — Robert H. Lurie Cancer Center
Locations (104):
- United States (104):
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Suburban Hospital, Bethesda, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin